CLINICAL TRIAL: NCT05283798
Title: Postpartum Intra-caesarean Section Insertion of Copper T380 Versus Multiload 375 IUD in a Randomized Controlled Trial.
Brief Title: Insertion of Copper T380 Versus Multiload IUD Post Partum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Abdelhameed Hussien Soliman (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Abdelhameed Hussien Soliman, resident, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: intra cs IUD
Record Dates: First submitted 2021-10-05; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-10

CONDITIONS: IUD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rate of missed threads in the first 6 weeks (Experimental): To compare efficacy safety & side effects of multiload 375 IUD versus copper T 380 IUD when inserted during elective CS
  Interventions: Device: IUD
- number of bleeding days in first 6 weeks (Other): compare numbers of bleeding days in first 6 weeks and first 6 month
  Interventions: Device: IUD

INTERVENTIONS:
Device: IUD — Postpartum intra-caesarean section insertion of copper T380 versus multiload 375

SUMMARY:
To compare efficacy safety & side effects of multiload 375 IUD versus copper T 380 IUD when inserted during elective CS

DETAILED DESCRIPTION:
Insertion of an intrauterine device (IUD) immediately after delivery is appealing for several reasons. The woman is known not to be pregnant, her motivation for contraception may be high, and the setting may be convenient for both the woman and her provider The World Health Organization (WHO) recommends that a woman should wait at least 24 months after delivery before the next pregnancy to decrease the adverse maternal, perinatal ,and infant outcomes.

Compared with other contraceptive methods, early post-partum IUD insertion has several advantages. It provides immediate contraception without interfering with breast feeding, and it may avoid discomfort related to insertion. Inserting an IUD immediately after placental removal has not been associated with increased infection, uterine perforation, postpartum bleeding, or uterine subinvolution . The expulsion rate is higher (approximately 12% in the first postpartum year) after immediate postpartum insertion compared to insertion 4 to 8 weeks later. Continuation rates are relatively high (87.6% and 76.3%, at 6 and 12 months, respectively Studies have shown that with effective provider training, the immediate postpartum IUD insertion (IPPIUD) complications such as expulsion, pelvic infection, bleeding, pain, missing threads ,and failure rates are not significantly different from those of interval PPIUD insertion (4:6 weeks) after delivery

ELIGIBILITY:
Inclusion Criteria:

women delivered by elective CS ≥ 36 wks

Exclusion Criteria:

Patients with PROM Patients on corticosteroids therapy Patients on anticoagulant patients who refuse participate in the study with written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all females in the reproductive age
Enrollment: 300 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
expulsion rate after 6 weeks of insertion | 6 weeks
  compare expulsion rates between the two types after 6 weeks by ultrasoud

SECONDARY OUTCOMES:
compare bleedind dayes and shift to anthor methoud | 6 weeks
  1. - number of bleeding days in the 1st 6 weeks
  2. - number of bleeding days in each month in the 1st 6 months
  3. compare by US between the 2 types
  4. - the shift into another method and what is it